CLINICAL TRIAL: NCT02457689
Title: A Randomized Phase I/II Study to Assess the Safety and Immunogenicity of the DNA-GTU Vaccine Administered by Two Novel Routes Compared to Placebo in HIV-infected Patients on Antiretroviral Therapy
Brief Title: The Safety and Immunogenicity of the DNA-GTU Vaccine Administered to HIV-infected Patients on ART vs Placebo
Acronym: CUTHIVTHER001
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 14SM2037
Record Dates: First submitted 2015-05-27; First posted 2015-05-29 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-10

CONDITIONS: HIV
Keywords: Human Immunodeficiency Virus; Immunodeficiency Virus, Human
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 (Transcutaneous and Placebo) (Placebo Comparator): Group 1 (Transcutaneous and Placebo) Participants will receive 1.0ml intramuscular injections of the vaccine Sodium Chloride BP into the upper thigh. Participants will also have a further 0.2ml of Sodium Chloride BP delivered transcutaneously. An area of skin of approximately 4 x 4cm will be photographed and prepared first. During this preparation, the area is shaved to remove the hair, and then superglue is applied to remove the top layer of skin (like waxing). The vaccine is spread onto the skin surface. Once applied, the area is covered with a comfeel bandage, the investigator will ask volunteers to not engage in strenuous exercise, shower, or bathe for 24 hours afterwards.
  Interventions: Other: Sodium chloride BP
- Group 2 (Transcutaneous and Active) (Active Comparator): Group 2 (Transcutaneous and Active) Participants will receive 1.0ml intramuscular injections of the GTU®-MultiHIV B Clade Vaccine (2 mg/ml) into the upper thigh. Participants will also have a further 0.2ml of the vaccine (2mg/ml) delivered transcutaneously. An area of skin of approximately 4 x 4cm will be photographed and prepared first. During this preparation, the area is shaved to remove the hair, and then superglue is applied to remove the top layer of skin (like waxing). The vaccine is spread onto the skin surface. Once applied, the area is covered with a comfeel bandage, the investigator will ask volunteers to not engage in strenuous exercise, shower, or bathe for 24 hours afterwards.
  Interventions: Biological: GTU®-MultiHIV B Clade Vaccine
- Group 3 (Electroporation and Placebo) (Placebo Comparator): Group 3 (Electroporation and Placebo) Participants will receive 1.0ml intramuscular injections of Sodium Chloride BP into the upper thigh using the ICHOR TriGridTM delivery system for intramuscular (TDS-IM) delivery with electroporation. Electroporation (EP) improves the delivery of the product into muscle cells, by delivering an electrical pulse with the injection using a hand held device that is pressed against your thigh. This will cause a muscle twitch with a sharp cramp-like feeling in the thigh lasting a few seconds. Once the procedure is carried out, the muscle will feel sore for up to 72 hours. The investigator will ask volunteers not to engage in any strenuous exercise for at least 24 hours after the procedure.
  Interventions: Other: Sodium chloride BP
- Group 4 (Electroporation and Active) (Active Comparator): Group 4 (Electroporation and Active) Participants will receive 1.0ml intramuscular injections of the GTU®-MultiHIV B Clade Vaccine (2mg/ml) into the upper thigh using the ICHOR TriGridTM delivery system for intramuscular (TDS-IM) delivery with electroporation. Electroporation (EP) improves the delivery of the product into muscle cells, by delivering an electrical pulse with the injection using a hand held device that is pressed against your thigh. This will cause a muscle twitch with a sharp cramp-like feeling in the thigh lasting a few seconds. Once the procedure is carried out, the muscle will feel sore for up to 72 hours. The investigator will ask volunteers not to engage in any strenuous exercise for at least 24 hours after the procedure.
  Interventions: Biological: GTU®-MultiHIV B Clade Vaccine

INTERVENTIONS:
Biological: GTU®-MultiHIV B Clade Vaccine — The investigational HIV-1 vaccine GTU®-MultiHIV B clade encodes for a MultiHIV antigen (synthetic fusion protein) built up by full-length polypeptides of Rev, Nef, Tat, p17 and p24 with more than 20 Th and CTL epitopes of protease, reverse transcriptase (RT) and gp160 regions of an HAN2 HIV-1 B clade isolate.
  Arms: Group 2 (Transcutaneous and Active); Group 4 (Electroporation and Active)
Other: Sodium chloride BP — For use in prophylactic and replacement therapy, requiring the use of isotonic saline solution.
  Arms: Group 1 (Transcutaneous and Placebo); Group 3 (Electroporation and Placebo)

SUMMARY:
CUT*HIVTHER 001 is a randomised placebo-controlled Phase I/II study aimed at exploring the safety and immunogenicity of two different modes of delivery of a GTU® DNA plasmid vaccine (GTU®-multiHIV B clade) in HIV infected volunteers on antiretroviral therapy (ART):

* Transcutaneous (TC) delivery to enhance intramuscular delivery and
* Electroporation (EP) enhanced intramuscular delivery Participants will be randomised 1:1:1 to TC:EP:saline for the purposes of analysis. Half the saline group will receive TC saline and half will receive EP saline.

  30 HIV infected male and female volunteers aged 18-45 years, who have been on ART for at least 6 months with 2 or more HIV plasma viral load measurements < 50 copies HIV RNA/ml prior to enrolment.

The investigational HIV-1 vaccine GTU®-MultiHIV B clade encodes for a MultiHIV antigen which is a synthetic fusion protein consisting of full-length polypeptides of Rev, Nef, Tat, p17 and p24 and containing more than 20 Th and CTL epitopes of protease, reverse transcriptase (RT) and gp160 regions of the HAN2 HIV-1 B clade.

Vaccine is provided in sealed vials at 2mg/ml, and a single 1ml IM injection of 2mg GTU®-MultiHIV DNA IM (into the thigh) is required to deliver a 2mg dose. Individuals in Group 2 will receive a further 0.4mg GTU®-MultiHIV DNA in 0.2ml administered by TC, a novel needle-free method of vaccine delivery.

DETAILED DESCRIPTION:
The investigators are exploring combination regimens with the overall aims of (i) optimising immune responses and (ii) developing safe and well tolerated strategies which will favour the development of T-cell responses that may enhance anti-HIV HIV therapy with the forward looking goal of working towards functional eradication of infection. The investigator proposes to combine the previously used IM and TC methods because preclinical data suggest that the combination of methods will favour the development of CD8 T cell responses. All groups will receive 6.0mg of the vaccine IM given in 3 doses over 12 weeks. Group 1 will receive the 6.0mg IM with electroporation (EP) and Group 2 will receive the 6.0mg IM without EP but together with an additional 1.2mg vaccine TC. The primary immunogenicity endpoint will be to determine whether either intervention group augments the cellular responses to vaccine specific peptides in relation to baseline. It is anticipated that none of subjects receiving saline placebo would have an increase in vaccine specific responses relative to those at baseline. Therefore if the differences between the active groups and saline placebo are sufficiently large, for example 80% responders in a GTU®-MultiHIV DNA active group, <10% in the control group, this would be significant.

Should the regimes prove safe, acceptable and induce significant immunogenicity then the intention is to move one or both regimes into a larger study powered to determine their potential long-term impact on therapy when used in combination with conventional ARV regimens. Proof of concept that DNA vaccination can induce de novo HIV specific responses that are associated with control of viral replication, would justify further investigation of their use in immunotherapies combined with ART intensification and/or anti-latency drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. Aged between 18 and 45 years on the day of screening
3. BMI between 19-30
4. Available for follow-up for the duration of the study
5. Willing and able to give written informed consent
6. HIV-1 Clade B infection documented by confirmed antibody test
7. Confirmed on 2 separate occasions in the 6 month period prior to enrolment to have viral load < 200 copies HIV RNA/ml whilst on ART
8. Nadir CD4+ > 250 CD4 lymphocytes AND screening CD4 >200 CD4 lymphocytes
9. Willing to avoid UV tanning or strong sun exposure during the immunisation period of the study
10. Willing to avoid all other vaccines within four weeks of scheduled study vaccinations
11. If heterosexually active female, using an effective method of contraception with partner (combined oral contraceptive pill; injectable or implanted contraceptive; consistent record with condoms if using these; physiological or anatomical sterility (in self or partner) from 14 days prior to the first vaccination until 4 months after the last, and willing to undergo urine pregnancy tests prior to each vaccination
12. If heterosexually active male, using an effective method of contraception with their partner from the first day of vaccination until 4 months after the last vaccination

Exclusion Criteria:

1. Pregnant or lactating
2. Use of regular topical treatment on the injection or application site within the last four weeks
3. UV tanning sessions or strong sun exposure within four weeks prior to enrolment
4. Excessive terminal hair growth on the investigational skin areas (to be assessed by reference to a photograph which will be available during screening visit)
5. Individuals in which a skin-fold measurement (cutaneous and subcutaneous tissue) of the upper right or left thigh exceeds 40 mm
6. Clinically relevant abnormality on history or examination including

   * history of grand-mal epilepsy, seizure disorder or any history of prior seizure
   * history of syncope or fainting episodes within 1 year of study entry
   * liver disease including active hepatitis B (surface antigen positive) or C (PCR positive)
   * any skin condition which may interfere with the trial assessment of the injection site
   * haematological, metabolic, gastrointestinal (excluding gastritis) or cardio-pulmonary disorders (excluding mild asthma)
   * a clinically significant abnormality on the ECG
   * autoimmune disease, or use of regular, systemic immunosuppressives in preceding 3 months
7. Known hypersensitivity to any component of the vaccine formulations used in this trial, or have severe or multiple allergies to drugs or pharmaceutical agents
8. History of severe local or general reaction to vaccination defined as

   1. local: extensive, indurated redness and swelling involving most of the antero-lateral thigh or the major circumference of the arm, not resolving within 72 hours
   2. general: fever >= 39.5oC within 48 hours; anaphylaxis; bronchospasm; laryngeal oedema; collapse; convulsions or encephalopathy within 72 hours
9. Receipt of live attenuated vaccine within 60 days of enrolment and any vaccine within 30 days of enrolment.
10. Receipt of an experimental vaccine containing HIV antigens at any time in the past
11. Receipt of immunoglobin within 4 months of screening
12. Participation in another trial of a medicinal product, completed less than 30 days prior to enrolment
13. Grade 2 or above routine laboratory parameters. Hyperbilirubinaemia to be considered an exclusion criterion only when confirmed to be conjugated bilirubinaemia
14. Current use of any electronic stimulation device, such as cardiac demand pacemakers, automatic implantable cardiac defibrillator, nerve stimulators, or deep brain stimulators.
15. Presence of any surgical or traumatic metal implants at the sites of administration
16. Unable to read and speak English to a fluency level adequate for the full comprehension of procedures required in participation and consent.
17. Unlikely to comply with protocol.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Grade 3 or above local solicited adverse event | Two weeks after final vaccination
Grade 3 or above systemic clinical and laboratory solicited adverse event | Four weeks after final vaccination
Any grade of adverse event that results in a clinical decision to discontinue further immunisations | Four weeks after final vaccination
Immunogenicity | Two weeks after final vaccination
  Change in IFN-γ ELISpot response to any of the pools of HIV-peptides encoded by the vaccine 2 weeks after the last immunisation relative to baseline, defined as a doubling in frequency from baseline or the presence of a response that was absent at baseline

SECONDARY OUTCOMES:
Any grade of adverse event that occurs in a participant that has received at least one immunisation | Two weeks after final vaccination
Immunogenicity | Two weeks after final vaccination
  Change in CD4+ and CD8+ T-cell cytokine responses (frequency and poly-functionality) to any of the pools of HIV peptides encoded by the vaccine, assessed by poly-chromatic ICS 2 weeks after the last immunisation

OTHER OUTCOMES:
Exploratory Immunogenicity | Four weeks after final vaccination
  Change from baseline in epitope recognition (frequency and magnitude) as determined by ELISpot analysis using overlapping 15mer peptides
Exploratory Immunogenicity | Four weeks after final vaccination
  Change from baseline in the magnitude of antigen-specific IgG Ab response
Exploratory Immunogenicity | Four weeks after final vaccination
  Change from baseline in HIV proviral DNA within PBMC
Exploratory Immunogenicity | Four weeks after final vaccination
  Change from baseline in HIV plasma viral load (number of copies of HIV RNA per millilitre), measured by quantitative PCR
Exploratory Immunogenicity | Four weeks after final vaccination
  Change from baseline in the immune activation and surface expression markers on T cells from baseline measured by poly-chromatic flow cytometry
Exploratory Immunogenicity | Four weeks after final vaccination
  Change from baseline in CD4+ lymphocyte count

CONTACTS AND LOCATIONS:
Overall Officials: Sheena McCormack, Phd, MD, Principal Investigator — Medical Research Council University College London
Locations (1):
- Imperial College London, Greater London, United Kingdom

REFERENCES:
- [Derived] Haidari G, Day S, Wood M, Ridgers H, Cope AV, Fleck S, Yan C, Reijonen K, Hannaman D, Spentzou A, Hayes P, Vogt A, Combadiere B, Cook A, McCormack S, Shattock RJ. The Safety and Immunogenicity of GTU(R)MultiHIV DNA Vaccine Delivered by Transcutaneous and Intramuscular Injection With or Without Electroporation in HIV-1 Positive Subjects on Suppressive ART. Front Immunol. 2019 Dec 13;10:2911. doi: 10.3389/fimmu.2019.02911. eCollection 2019. PMID 31921170